CLINICAL TRIAL: NCT06064942
Title: Multiple Family Narrative Therapy as Treatment for Chinese Families of Children With Attention-Deficit/Hyperactivity Disorder: A Randomised Controlled Trial
Brief Title: Multiple Family Narrative Therapy for Chinese Families of Children With Attention Deficit Hyperactivity Disorder
Acronym: MFNT-CADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: University Grants Committee, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGC Ref No. 12615322; General Research Fund (GRF) (Other Grant/Funding Number: University Grants Committee (UGC))
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-04

CONDITIONS: Attention-deficit/Hyperactivity Disorder; Special Education; Special Needs Children; Attention Deficit Disorder; Hyperactivity Disorder
Keywords: Attention deficit; Hyperactivity disorder; Multiple family group; Narrative therapy; Efficacy; Special educational needs; Intervention; Parent-child
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFNT Intervention (Treatment Group) (Experimental): Parents of children with ADHD who are randomized in Treatment Group will first take part in a pre-tested 4-session MFNT intervention programme. The parents will participate in lectures, group discussions, video demonstrations, and in-group exercises offered in these four mentored sessions, while their children will attend the second and fourth sessions.
  Interventions: Behavioral: Multiple Family Narrative Therapy (MFNT)
- MFNT Intervention (Wait Listing Control Group) (Experimental): Families of children with ADHD who are randomized in Wait Listing Control Group receive services as usual by the school social personnel during the intervention period. The 4-session MFNT intervention program will be delivered to them after the intervention period.
  Interventions: Behavioral: School services for families of children with ADHD

INTERVENTIONS:
Behavioral: Multiple Family Narrative Therapy (MFNT) — MFNT consist of 4 weekly group sessions with selected themes from both multiple family therapy (MFT) and narrative therapy (NT) offered in a group format. Parents participates in four mentored sessions, while their children attend the second and fourth sessions. The family is treated as a system through both psychodynamic practices and attachment theories to manage symptoms, to achieve family resilience, and to empower both parents and child to share their unique and lived value-driven experiences. MFNT provides families with therapeutic environments that are conducive to learning and modelling in order to facilitate the process of building healthier parent-child dyads.
  Arms: MFNT Intervention (Treatment Group)
Behavioral: School services for families of children with ADHD — Selected school social personnel will deliver services as usual for the control group.
  Arms: MFNT Intervention (Wait Listing Control Group)

SUMMARY:
The goal of this randomized controlled trial is to develop and to implement a multiple family narrative therapy intervention consisting of parent-child relationships training among Chinese families of children with attention deficit hyperactivity disorder (ADHD). The intervention aims to reduce the psychological distress of parents and their child, thus improving parent-child relationships, and the trial aims to assess the effectiveness of MFNT among them. A RCT design supplemented by qualitative interviews will be used to evaluate the effectiveness of multiple family narrative therapy intervention on family welfare.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) affects 6.4% of children in Hong Kong while medicating children with ADHD in Hong Kong has increased 36-fold between 2001 and 2015. Global studies provide evidence that children with ADHD have experienced a substantial amount of stress due to the childrearing distress of their parents. The education system in Hong Kong is exceptionally competitive and academically focused. When parenting skills are measured against the academic achievement of children, parents may feel helpless and hopeless, which contribute to social isolation during stressful times that stem from caring for a child with ADHD or other developmental disabilities. Chinese parents who are heavily burdened by the pressure of preventing the academic failure of their children typically resort to outing their children in privately operated tutorial classes and giving them additional home-based assignments. These remedial actions often increase the stress levels of both parents and child. In the Chinese culture, academic failure shames the family, which leads to parent-child conflicts and mental health issues. These family problems can negatively affect Chinese children with ADHD.

Related support services in Hong Kong are also inadequate and insufficient. The management of ADHD in Hong Kong follows the international mainstream treatments that comprise prescribing stimulant medication and behavioural interventions. Few studies on psychoeducation models have focused on parent-child relationships, parental stress for families of children with learning disabilities in Hong Kong. The available psychological approaches mainly address the behavioural changes of children with special educational needs (SENs). However, the psychoeducation approach does not reduce the social isolation of parents and the stigmatisation of medication by parents who fear the side effects and long-term effects. To address this research gap, a psychotherapy model is used to evaluate the impact of its intervention on both parents and their child with SENs, especially ADHD, which has been recently seen an increase in demand. At the same time, it is crucial to examine the process of change in attitudes and interactions among family members who participate in Multiple Family Narrative Therapy (MFNT) so that helping professionals can learn from this qualitative part to refine the design and session plan of MFNT.

This study addresses a need in the Hong Kong Chinese community with four anticipated outcomes: 1) the effectiveness of MFNT as a brief-targeted intervention model with CFCAs is determined; 2) a participatory approach that engages both parents and children is realised; 3) a culturally applicable practice manual for the Chinese context is produced; and 4) the use of the practice manual by school and integrative family services is encouraged.

This study evidence-informed and knowledge-building results will support a brief-targeted MFNT approach in Hong Kong to supplement the "treatment as usual" school-focused process in working with Chinese families of children with ADHD (CFCAs) towards a collaborative model where family members can reassess their identity and adopt alternative interaction behaviours. Excessive school-based work increases the pressure of students in an academic achievement-driven culture, which intensifies conflicts in parent-child relationships.

A randomized controlled trial (RCT) design and qualitative interviews will be used to evaluate the effectiveness of MFNT on family welfare. The first objective is to examine the effectiveness of a brief-targeted MFNT for CFCAs in Hong Kong. The aim is to reduce their psychological distress to enhance parent-child relationships. The second objective is to assess and document the course of change in attitudes and interactions among the MFNT participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants 7-13 years old and their parents
* ADHD diagnosis (by psychiatrist or educational psychologist)
* Diagnosis with comorbidity of other learning disabilities
* Cantonese speaking participants (child and parents)
* At least one of the parents, but not siblings nor grandparents, can commit to all four sessions
* Participants able to comply with all testing and study requirements

Exclusion Criteria:

* Formal current diagnosis of psychosis
* Limitation in daily communication
* Previous service recipients of Narrative Therapy or Multiple Family Group
* Non-Cantonese speaking child or parent
* Parents or children who refuse to give written consent for their participation in the study

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Kessler Psychological Distress Scale (KPDS) | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  Kessler Psychological Distress Scale is a 10-item scale completed by the child and the child's parent. It assesses the frequency of distress-related feelings in the past month on a 5-point Likert Scale (1=None of the time; 2=A little of the time; 3=Some of the time; 4=Most of the time; 5=All of the time). The scale is reliable and valid for the local context, given it will be delivered in Chinese. Changes in scores of Kessler Psychological Distress Scale will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Parental Stress Scale (PSS) | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  Parental Stress Scale (PSS) consists of 17 items on a 6-point scale (1 = strongly disagree; 2 = disagree; 3= somewhat disagree; 4 = somewhat agree; 5 = agree; 6 = strongly agree) measuring parents' perception of parental stress. Seven items require reverse scoring. A total score is calculated, with higher scores indicating higher levels of parental stress. The Chinese version of the scale has been translated and validated. Changes in its total score will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Parent-Child Relationship Scale | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  Parent-Child Relationship Scale is a scale that assesses subjects' perceptions of their current relationship with their children. It consists of 17 items based on 5-point scale, ranging from 1 = never to 5 = always. The scale uses mean score, and a higher score indicates a more positive parent-child relationship. Changes in its mean score will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Parental Acceptance-Rejection Questionnaire (PARQ) | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  The Parental Acceptance-Rejection Questionnaire (PARQ) is a self-report instrument designed to measure individuals' perceptions of parental acceptance-rejection. It consisted of four scales: (1) warmth/affection, (2) hostility/aggression, (3) indifference/neglect, and (4) undifferentiated rejection. The child version assesses children's current perceptions of the degree to which they experienced parental (maternal and paternal) acceptance or rejection in childhood, and it is suitable for children older than 7 years. The parent version asks parents to assess the way they now treat their children. Both scales are rated on 4-point Likert scale (Almost Never True = 1, Rarely True = 2, Sometimes True = 3, Almost Always True = 4) Changes in the scores of subscales namely (1) warmth/affection, (2) hostility/aggression, (3) indifference/neglect, and (4) undifferentiated rejection in both father and mother will be evaluated before, after the intervention.
Parental Bonding Inventory (PBI) | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  Parental Bonding Inventory (PBI) is a 25-item instrument assessing levels of parental care and overprotection perceived by the child. It consisted of two subscales termed 'care' and 'overprotection/control'. The measure is to be completed for both mothers and fathers separately, with each parent being scored on a 4-point Likert scale (Very unlike = 0, Moderately unlike = 1, Moderately like = 2, Very like = 3). Changes in the scores in "care" and "overprotection/control" subscales in both father and mother will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).

SECONDARY OUTCOMES:
Satisfaction With Family Life Scale (SWFL) | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  Satisfaction With Family Life Scale (SWFL) is a 5-item scale that assesses an individual's global judgment of family satisfaction. Parents and children were required to agree or disagree with global statements about family life on a 7-point Likert-type scale ranging from 1 = strongly disagree to 7 = strongly agree. This instrument has been successfully used in a variety of family samples and offers a brief, widely applicable tool to measure satisfaction with family life. Changes in its total score will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Guilt and Shame Questionnaire (GSQ) | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  Guilt and Shame Questionnaire (GSQ) is a 10-item scale to assess one's feelings of guilt and shame associated with disabilities including but not limited to mental illness. It consisted of two subscale - shame and guilt, both are rated on a 5-point Likert scale ranging from 1 (never) to 5 (always). The scale was completed by parents and children. The evaluation of guilt and shame is calculated based on the sum scores of each subscale. Changes in scores of total scale, guilt and shame subscales will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention).
Walsh Family Resilience Questionnaire (WFRQ) | 1-week prior intervention, Intervention week 4, and 3 months post-intervention
  Walsh Family Resilience Questionnaire (WFRQ) is a scale that assesses to what extent individual statements are truthful about how their family is coping with crises and ongoing challenges. The WFRQ consists of three main scales: belief systems (10 items), organisation, communication and problem-solving (13 items), and utilizing external resources (3 items). The scale asked the parents to complete on a 5-point scale (Rarely/Never= 1, Not Often= 2, Sometimes= 3, Often= 4, Almost Always= 5) Changes in the scores of subscales of (1) belief systems and (2) organisation, communication and problem-solving will be evaluated before, after the intervention as well as at a follow-up assessment (3 months after the end of the intervention). The subscale namely "utilizing external resources" was not included in the study as this dimension is conceptually irrelevant to the intervention process.

CONTACTS AND LOCATIONS:
Overall Officials: Tak Mau Chan, PhD, Principal Investigator — Hong Kong Baptist University
Locations (1):
- Department of Social Work, Hong Kong Baptist University, Hong Kong, China, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided